CLINICAL TRIAL: NCT02050087
Title: The Role of Postoperative Immobilization After Arthroscopic Rotator Cuff Repair: A Prospective Randomized Controlled Non-inferiority Trial
Brief Title: The Role of Postoperative Immobilization After Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lovisenberg Diakonale Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/2288
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Rotator Cuff Rupture
Keywords: Rotator cuff; Rehabilitation
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 weeks with simple sling (Active Comparator): Early motion after arthroscopic rotator cuff repair.
  Interventions: Device: Neutral brace
- 6 weeks with neutral brace (Active Comparator): Delayed motion after arthroscopic rotator cuff repair.
  Interventions: Device: Simple sling.

INTERVENTIONS:
Device: Simple sling.
  Arms: 6 weeks with neutral brace
Device: Neutral brace
  Arms: 3 weeks with simple sling

SUMMARY:
The study is a prospective randomized controlled non-inferiority trial where we elucidate the role of postoperative immobilization after arthroscopic rotator cuff repair.

DETAILED DESCRIPTION:
Rotator cuff tendon injury ranks among the most prevalent of shoulder disorders causing pain and impaired function, and is a major socioeconomic burden on society. The study is a prospective randomized controlled non-inferiority trial where we elucidate the role of postoperative immobilization after arthroscopic rotator cuff repair. Our primary goal is to compare clinical and structural results after rotator cuff repair and to compare a restrictive and an active postoperative rehabilitation protocol. Our secondary goal is to establish guidelines for optimized rehabilitation after rotator cuff repair to ensure the best possible outcome for this large group of patients. Our aim is also to establish guidelines for timing of return to work. The major complications following rotator cuff repair and the current rehabilitation regimens are rotator cuff retears and postoperative stiffness. The information obtained in this study may enable development of targeted, cost-effective treatment and rehabilitation with good, lasting long-term results.

ELIGIBILITY:
Inclusion Criteria: Repairable partial- or full-thickness rotator cuff tear affecting supraspinatus and/or upper infraspinatus tendon -

Exclusion Criteria: Irreparable or incomplete repairable tears of supraspinatus and/or infraspinatus tendon.

Large/massive rotator cuff tear. Diabetes mellitus. Systemic inflammatory disorder. Fatty muscle infiltration >grade 2 (Goutallier). Subscapularis tendon tear. Adhesive capsulitis. Concomitant labral repair. Revision repair.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
We define Western Ontario Rotator Cuff (WORC) index at 12 months after surgery as the primary endpoint | One year
  We define Western Ontario Rotator Cuff (WORC) index at 12 months after surgery as the primary endpoint. We will compare WORC of the early range of motion group to a delayed range of motion group.

CONTACTS AND LOCATIONS:
Overall Officials: Sigbjørn Dimmen, MD, Phd, Study Chair — Lovisenberg Diaconal Hospital, Oslo, Norway
Locations (1):
- Lovisenberg Diaconal Hospital, Oslo, Norway